CLINICAL TRIAL: NCT06398236
Title: Multicentre, Exploratory, Prospective, Open-labelled, Non-controlled Study to Evaluate the Effect of SE5-OH Tablets on Healthy Women With Menopausal Symptoms
Brief Title: Open-labelled Study to Evaluate the Effect of SE5-OH Tablets on Healthy Women With Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrition & Sante Iberia (Industry)
Collaborators: Adknoma Health Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EQUELLE_22_01
Record Dates: First submitted 2024-04-09; First posted 2024-05-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Menopause
MeSH Terms: interventions — SE5-OH

STUDY DESIGN:
Intervention Model Description: Multicentre, exploratory, prospective, open-labelled study to evaluate the efficacy of SE5-OH tablets on menopausal symptoms in healthy women experiencing menopausal symptoms after 12 weeks of administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SE5-OH tablets (Experimental): The product under investigation is a food supplement that contains SE5-OH (Fermented Soy germ, include S-equol), Crystalline cellulose, Oats fiber, Agar, Cyclic oligosaccharide, HPMC, Reduced syrup. The food supplement is presented in sealed bottles, each bottle contains 120 tablets with the recommended daily dose of 4 tablets per day administrated orally with a glass of water. The 4 tablets can be administrated together in a unique intake or in 2 separated intakes (2 tablets/intake) along the day.
  Interventions: Dietary Supplement: SE5-OH tablets

INTERVENTIONS:
Dietary Supplement: SE5-OH tablets — SE5-OH (Fermented Soy germ, include S-equol), Crystalline cellulose, Oats fiber, Agar, Cyclic oligosaccharide, HPMC, Reduced syrup.

SUMMARY:
Multicentre, exploratory, prospective, open-labelled study to evaluate the efficacy of SE5-OH tablets on menopausal symptoms in healthy women experiencing menopausal symptoms after 12 weeks of administration.

The study will be performed in 10 hospitals (private and public) located in Spain. Recruitment period of 6 months will be defined in order to include up to 300 healthy volunteers from different national hospitals and clinics.

DETAILED DESCRIPTION:
Multicentre, exploratory, prospective, open-labelled, non-controlled study to evaluate the efficacy of SE5-OH tablets for menopausal symptoms reduction. SE5-OH tablets are a food supplement containing active S-equol. The daily dose of S-equol is 10 mg in the form of 4 tablets of SE5-OH tablets.

The study will be performed in 10 hospitals (private and public) located in Spain to include up to 300 subjects in 6 months of recruitment period.

Investigators will review the medical history from healthy women with moderate to severe menopausal symptoms who are visiting the participating site, investigators will ensure that each candidate meets all the inclusion criteria and none of exclusion criteria. Suitable participants will be informed during the visit about the nature of the investigational study by receiving first information about the investigational product (food supplement) and invited to participate later when all questions have been addressed. A 14 days' period of reflexion is possible for every participant in accordance with Good Clinical Practice.

The procedures involved will be explained in detail and written consent must be obtained with subject and investigators signature before subject participation. The total duration of each participant in the study will be 16 weeks (12 weeks treatment + 4 weeks follow up). The participation in the study is completely voluntary.

The study consists of 4 visits: 3 visits until the end of treatment (EoT) with 1 follow up/end of study visit (FU/EoS) after treatment completion.

SE5-OH tablets will be administrated in tablets (4 per day) by daily oral intake until the day before the end of treatment date (week 12). Non-administrated SE5-OH tablets and VMS diary competition will be verified during the study in the corresponding visits until the EoS (visit 4).

ELIGIBILITY:
Inclusion Criteria:

* 45-60 years healthy women who have provided signed ICF.
* Experiencing menopause symptoms for at least 1 month.
* Total MRS score ≥9 at inclusion time (baseline).

MRS with a score equal or above 9 include women with moderate to severe menopausal symptoms according to the validated analysis of this questionnaire.

Exclusion Criteria:

* Women currently receiving hormone replacement therapy (HRT) or bio identical hormone replacement therapy (BHRT) or have received HRT/BHRT in the last 3 months.
* Pregnant, nursing women or women planning to become pregnant*.
* Subject with a history or presence of clinically severe disease such as hepatic, renal, endocrine, hematologic, immunologic (including chronic inflammatory conditions) and cancer disease.
* History or presence psychosomatic diseases (drug treatment), epilepsy, rheumatism.
* Allergies to soy.
* History of any food behaviour complication (lacking sufficient intake and/or over intake of food)
* Intestinal malabsorption that could decrease food supplements intestinal absorption.
* Receiving any drug during the last 3 months for menopause symptoms or any food supplement during the last 1 month that could decrease or hide/mask the effect of the experimental product.
* Participation to another clinical trial.
* Any other medical problem identified by the investigator that could alter the ability of the volunteer to participate to the study including non-treated/non controlled thyroid disease, diabetes (among others).

  * A negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or HCG equivalent units) must be performed prior to subject enrolment and must be negative 24 hours prior to initiation of study treatment in case of any suspicious.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of SE5-OH tablets on menopausal symptoms. | At week 12 from week 0.
  To evaluate the efficacy of SE5-OH tablets on menopausal symptoms with the assessment of the menopausal rating scale (MRS) total scores and subscales scores (somatic, psychological, and urogenital) after 12 weeks of treatment from week 0.
  MRS consists of a list of 11 symptoms, that can get 0 (no symptom) or up to 4 scoring points (severe symptom) depending on the severity of the complaints perceived by the women completing the scale.
  The total score of the MRS ranges between 0 (asymptomatic) and 44 (highest degree of complaints) and is the sum of the dimension scores. The total score can be categorized into: No little (0-4) / Mild (5-8) / Moderate (9-15) / Severe (≥16).
  Higher scores mean worse outcome.

SECONDARY OUTCOMES:
To evaluate the changes in menopausal symptoms. | At week 4 and 16 from week 0.
  To evaluate the changes in menopausal symptoms by MRS total scores and subscales scores (somatic, psychological, and urogenital) at week 4 and 16 from week 0.
  MRS consists of a list of 11 symptoms, that can get 0 (no symptom) or up to 4 scoring points (severe symptom) depending on the severity of the complaints perceived by the women completing the scale.
  The total score of the MRS ranges between 0 (asymptomatic) and 44 (highest degree of complaints) and is the sum of the dimension scores. The total score can be categorized into: No little (0-4) / Mild (5-8) / Moderate (9-15) / Severe (≥16).
  Higher scores mean worse outcome.
To evaluate the changes in vulvovaginal symptoms. | At week 4, 12 and 16 from week 0.
  To evaluate the changes in vulvovaginal symptoms by the vulvovaginal symptoms questionnaire (VSQ) total score and subscales score (symptoms, emotions, life-impact, and sexual impact) at week 4, 12 and 16 from week 0.
  VSQ consists of a list of 21 items answered as yes (1 point) or no (0 points), and making up a total of four scales:
  * Vulvovaginal symptoms: 0 to 7 points (items 1-7)
  * Emotions: 0 to 4 points (items 8-11)
  * Life-impact: 0 to 4 points (items 12-15)
  * Sexual impact: 0 to 5 points (items 16, 18-21) [item 17 asks about sexual activity, if the answer is affirmative then the four scales are evaluated, if it is negative, only the first three] The total score of the VSQ ranges between 0 and 20: the higher the score, the worse the rating
To evaluate the changes in work performance associated to menopausal symptoms. | At week 12 from week 0.
  To evaluate the changes in work performance associated to menopausal symptoms, the utrecht work engagement scale (UWES) total scores and subscales scores (vigor, dedication, and absorption) at week 12 from week 0.
  UWES consists of a list of 17 items, that can get 0 (never) or up to 6 scoring points (always / every day). There are 3 scales:
  * Vigor (item 1, 4, 8, 12, 15, 17)
  * Dedication (item 2, 5, 7, 10, 13)
  * Absorption (item 3, 6, 9, 11, 14, 16) The mean scale score of the three UWES subscales is computed by adding the scores on the particular scale and dividing the sum by the number of items of the subscale involved. A similar procedure if followed for the total score. Hence, the UWES, yields three subscale scores and/or a total score that range between 0 and 6: the higher score, the most work engagement.
To evaluate the changes in pain in joint and hand, shoulder, and low back. | At week 12 from week 0
  To evaluate the changes in pain in joint and hand, shoulder, and low back by the visual analogue scale (VAS) at week 12 from week 0. Each visual analogue scale scores from 0 to 10. Higher scores mean worse outcome.
To evaluate the changes in sleep quality. | At week 12 from week 0.
  To evaluate the changes in sleep quality by the visual analogue scale (VAS) at week 12 from week 0.
  Visual analogue scale scores from 0 to 10. Higher scores mean worse outcome.
To evaluate the changes in vasomotor symptoms. | At week 4, 12 and 16 from week 0 based on daily registrations.
  To evaluate the changes in vasomotor symptoms (VMS) such hot flushes and night sweats, a registration of frequency and severity every day during the 16 weeks of subject participation.
  The mean number of hot flashes/night sweats by severity (mild, moderate, and severe) reported in the diary will be calculated in each study period.
To evaluate the changes in the vaginal maturation index. | At week 4, 12 and 16 from week 0.
  To evaluate the changes in the vaginal maturation index (VMI) by pap smear at week 4, 12 and 16 from week 0.
  The VMI is presented as 0/0/0, representing respectively: % parabasal cells, % intermediate cells and % superficial cells.
  The VMI is the ratio of different cell types in the vaginal wall (parabasal, intermediate and superficial cells) the presence of one and another type is influenced by oestrogen and progesterone stimulation, which means, that VMI will change throughout a woman's life depending on age and/or reproductive stage. Vaginal pH >5 seems to be associated to dryness and mucosal pallor; hormonal changes could affect either to vaginal pH and vaginal epithelium resulting in signs and symptoms of dryness or dyspareunia among others. Weber et al. concluded in their study that objective assessments such VMI and vaginal pH should be evaluated in conjunction with subjective assessments.
To evaluate the changes in the vaginal pH. | At week 4, 12 and 16 from week 0.
  To evaluate the changes in the vaginal pH (VpH) by a pH determination at week 4, 12 and 16 from week 0.
To evaluate the changes in body mass index (BMI). | At week 12 from week 0.
  To evaluate the changes in body mass index (BMI) at week 12 from week 0. Weight and height will be combined to report BMI in kg/m^2
To evaluate the changes in blood pressure (BP). | At week 16
  To evaluate the changes in blood pressure (BP) at week 12 from week 0. Systolic and Diastolic Blood Pressure will be reported in mmHg.
To evaluate the variability of equol producers and equol non-producers among the subjects. | At week 16
  Equol producers vs non-equol producers will be described at week 16 by means of results from urine analysis:
  * S-equol concentration
  * Daidzein concentration
  * S-equol/daidzein Log10 The patients will be classified into equol producer / non-producer / indeterminate, considering that daidzein ratio of -1.75 provided a demarcation to define equol producer status.
To evaluate the adverse events. | Up to 16 weeks.
  Adverse events (in terms of severity, intensity, causal relationship and outcome) will be assessed during the 16 weeks of study participation.
To evaluate tolerability. | At week 16
  The perception of tolerability by subject and investigator will be described at week 16. It will be measured with the folowing scale: excelent/good/moderate/poor/not evaluated by each one of them.
To evaluate the compliance. | At week 12
  Compliance (in terms of poor, moderate good and very good) during the 12 weeks of treatment administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Palacios Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Background] Goodman NF, Cobin RH, Ginzburg SB, Katz IA, Woode DE; American Association of Clinical Endocrinologists. American Association of Clinical Endocrinologists Medical Guidelines for Clinical Practice for the diagnosis and treatment of menopause. Endocr Pract. 2011 Nov-Dec;17 Suppl 6:1-25. doi: 10.4158/ep.17.s6.1. No abstract available. PMID 22193047
- [Background] Portman DJ, Gass ML; Vulvovaginal Atrophy Terminology Consensus Conference Panel. Genitourinary syndrome of menopause: new terminology for vulvovaginal atrophy from the International Society for the Study of Women's Sexual Health and The North American Menopause Society. Climacteric. 2014 Oct;17(5):557-63. doi: 10.3109/13697137.2014.946279. Epub 2014 Aug 25. PMID 25153131
- [Background] Brimacombe J, Berry A. The laryngeal mask airway for dental surgery--a review. Aust Dent J. 1995 Feb;40(1):10-4. doi: 10.1111/j.1834-7819.1995.tb05605.x. PMID 7710408
- [Background] Delamater L, Santoro N. Management of the Perimenopause. Clin Obstet Gynecol. 2018 Sep;61(3):419-432. doi: 10.1097/GRF.0000000000000389. PMID 29952797
- [Background] Avis NE, Stellato R, Crawford S, Bromberger J, Ganz P, Cain V, Kagawa-Singer M. Is there a menopausal syndrome? Menopausal status and symptoms across racial/ethnic groups. Soc Sci Med. 2001 Feb;52(3):345-56. doi: 10.1016/s0277-9536(00)00147-7. PMID 11330770
- [Background] Couzi RJ, Helzlsouer KJ, Fetting JH. Prevalence of menopausal symptoms among women with a history of breast cancer and attitudes toward estrogen replacement therapy. J Clin Oncol. 1995 Nov;13(11):2737-44. doi: 10.1200/JCO.1995.13.11.2737. PMID 7595732
- [Background] Palacios S, Stevenson JC, Schaudig K, Lukasiewicz M, Graziottin A. Hormone therapy for first-line management of menopausal symptoms: Practical recommendations. Womens Health (Lond). 2019 Jan-Dec;15:1745506519864009. doi: 10.1177/1745506519864009. PMID 31378196
- [Background] Marjoribanks J, Farquhar C, Roberts H, Lethaby A, Lee J. Long-term hormone therapy for perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2017 Jan 17;1(1):CD004143. doi: 10.1002/14651858.CD004143.pub5. PMID 28093732
- [Background] Nappi RE, Kroll R, Siddiqui E, Stoykova B, Rea C, Gemmen E, Schultz NM. Global cross-sectional survey of women with vasomotor symptoms associated with menopause: prevalence and quality of life burden. Menopause. 2021 May 24;28(8):875-882. doi: 10.1097/GME.0000000000001793. PMID 34033602
- [Background] Krizova L, Dadakova K, Kasparovska J, Kasparovsky T. Isoflavones. Molecules. 2019 Mar 19;24(6):1076. doi: 10.3390/molecules24061076. PMID 30893792
- [Background] Setchell KD, Clerici C. Equol: history, chemistry, and formation. J Nutr. 2010 Jul;140(7):1355S-62S. doi: 10.3945/jn.109.119776. Epub 2010 Jun 2. PMID 20519412
- [Background] Mayo B, Vazquez L, Florez AB. Equol: A Bacterial Metabolite from The Daidzein Isoflavone and Its Presumed Beneficial Health Effects. Nutrients. 2019 Sep 16;11(9):2231. doi: 10.3390/nu11092231. PMID 31527435
- [Background] Weber MA, Limpens J, Roovers JP. Assessment of vaginal atrophy: a review. Int Urogynecol J. 2015 Jan;26(1):15-28. doi: 10.1007/s00192-014-2464-0. Epub 2014 Jul 22. PMID 25047897
- [Background] Messina M, Nagata C, Wu AH. Estimated Asian adult soy protein and isoflavone intakes. Nutr Cancer. 2006;55(1):1-12. doi: 10.1207/s15327914nc5501_1. PMID 16965235
- [Background] Setchell KD, Clerici C, Lephart ED, Cole SJ, Heenan C, Castellani D, Wolfe BE, Nechemias-Zimmer L, Brown NM, Lund TD, Handa RJ, Heubi JE. S-equol, a potent ligand for estrogen receptor beta, is the exclusive enantiomeric form of the soy isoflavone metabolite produced by human intestinal bacterial flora. Am J Clin Nutr. 2005 May;81(5):1072-9. doi: 10.1093/ajcn/81.5.1072. PMID 15883431
- [Background] Khatoon A, Husain S, Husain S, Hussain S. An Overview of Menopausal Symptoms Using the Menopause Rating Scale in a Tertiary Care Center. J Midlife Health. 2018 Jul-Sep;9(3):150-154. doi: 10.4103/jmh.JMH_31_18. PMID 30294188
- [Background] Ahsan M, Mallick AK. The Effect of Soy Isoflavones on the Menopause Rating Scale Scoring in Perimenopausal and Postmenopausal Women: A Pilot Study. J Clin Diagn Res. 2017 Sep;11(9):FC13-FC16. doi: 10.7860/JCDR/2017/26034.10654. Epub 2017 Sep 1. PMID 29207728
- [Background] Erekson EA, Yip SO, Wedderburn TS, Martin DK, Li FY, Choi JN, Kenton KS, Fried TR. The Vulvovaginal Symptoms Questionnaire: a questionnaire for measuring vulvovaginal symptoms in postmenopausal women. Menopause. 2013 Sep;20(9):973-9. doi: 10.1097/GME.0b013e318282600b. PMID 23481118
- [Background] Fong TC, Ng SM. Measuring engagement at work: validation of the Chinese version of the Utrecht Work Engagement Scale. Int J Behav Med. 2012 Sep;19(3):391-7. doi: 10.1007/s12529-011-9173-6. PMID 21681564
- [Background] Alqurashi YD, Dawidziuk A, Alqarni A, Kelly J, Moss J, Polkey MI, Morrell MJ. A visual analog scale for the assessment of mild sleepiness in patients with obstructive sleep apnea and healthy participants. Ann Thorac Med. 2021 Apr-Jun;16(2):141-147. doi: 10.4103/atm.ATM_437_20. Epub 2021 Feb 19. PMID 34012480
- [Background] Thurston RC, Joffe H. Vasomotor symptoms and menopause: findings from the Study of Women's Health across the Nation. Obstet Gynecol Clin North Am. 2011 Sep;38(3):489-501. doi: 10.1016/j.ogc.2011.05.006. PMID 21961716
- [Background] Gold EB, Colvin A, Avis N, Bromberger J, Greendale GA, Powell L, Sternfeld B, Matthews K. Longitudinal analysis of the association between vasomotor symptoms and race/ethnicity across the menopausal transition: study of women's health across the nation. Am J Public Health. 2006 Jul;96(7):1226-35. doi: 10.2105/AJPH.2005.066936. Epub 2006 May 30. PMID 16735636
- [Background] Nappi RE, Martini E, Cucinella L, Martella S, Tiranini L, Inzoli A, Brambilla E, Bosoni D, Cassani C, Gardella B. Addressing Vulvovaginal Atrophy (VVA)/Genitourinary Syndrome of Menopause (GSM) for Healthy Aging in Women. Front Endocrinol (Lausanne). 2019 Aug 21;10:561. doi: 10.3389/fendo.2019.00561. eCollection 2019. PMID 31496993
- [Background] Society of Obstetricians and Gynaecologists of Canada. SOGC clinical practice guidelines. The detection and management of vaginal atrophy. Number 145, May 2004. Int J Gynaecol Obstet. 2005 Feb;88(2):222-8. doi: 10.1016/j.ijgo.2004.11.003. PMID 15779109
- [Background] Sathyapalan T, Aye M, Rigby AS, Thatcher NJ, Dargham SR, Kilpatrick ES, Atkin SL. Soy isoflavones improve cardiovascular disease risk markers in women during the early menopause. Nutr Metab Cardiovasc Dis. 2018 Jul;28(7):691-697. doi: 10.1016/j.numecd.2018.03.007. Epub 2018 Apr 10. PMID 29739677
- [Background] Linderman GC, Lu J, Lu Y, Sun X, Xu W, Nasir K, Schulz W, Jiang L, Krumholz HM. Association of Body Mass Index With Blood Pressure Among 1.7 Million Chinese Adults. JAMA Netw Open. 2018 Aug 3;1(4):e181271. doi: 10.1001/jamanetworkopen.2018.1271. PMID 30646115
- [Background] Taku K, Melby MK, Kronenberg F, Kurzer MS, Messina M. Extracted or synthesized soybean isoflavones reduce menopausal hot flash frequency and severity: systematic review and meta-analysis of randomized controlled trials. Menopause. 2012 Jul;19(7):776-90. doi: 10.1097/gme.0b013e3182410159. PMID 22433977
- [Background] Colacurci N, De Franciscis P, Atlante M, Mancino P, Monti M, Volpini G, Benvenuti C. Endometrial, breast and liver safety of soy isoflavones plus Lactobacillus sporogenes in post-menopausal women. Gynecol Endocrinol. 2013 Mar;29(3):209-12. doi: 10.3109/09513590.2012.738724. Epub 2012 Nov 30. PMID 23194023
- [Background] Alekel DL, Genschel U, Koehler KJ, Hofmann H, Van Loan MD, Beer BS, Hanson LN, Peterson CT, Kurzer MS. Soy Isoflavones for Reducing Bone Loss Study: effects of a 3-year trial on hormones, adverse events, and endometrial thickness in postmenopausal women. Menopause. 2015 Feb;22(2):185-97. doi: 10.1097/GME.0000000000000280. PMID 25003624
- [Background] Nahas EA, Nahas-Neto J, Orsatti FL, Carvalho EP, Oliveira ML, Dias R. Efficacy and safety of a soy isoflavone extract in postmenopausal women: a randomized, double-blind, and placebo-controlled study. Maturitas. 2007 Nov 20;58(3):249-58. doi: 10.1016/j.maturitas.2007.08.012. Epub 2007 Oct 29. PMID 17913408
- [Background] Palacios S, Pornel B, Vazquez F, Aubert L, Chantre P, Mares P. Long-term endometrial and breast safety of a specific, standardized soy extract. Climacteric. 2010 Aug;13(4):368-75. doi: 10.3109/13697131003660585. PMID 20380569
- [Background] Messina M. The endometrial effects of isoflavones: a discussion paper. Complement Ther Clin Pract. 2008 Aug;14(3):212-4. doi: 10.1016/j.ctcp.2008.04.005. Epub 2008 Jun 20. No abstract available. PMID 18640633
- [Background] Hooper L, Madhavan G, Tice JA, Leinster SJ, Cassidy A. Effects of isoflavones on breast density in pre- and post-menopausal women: a systematic review and meta-analysis of randomized controlled trials. Hum Reprod Update. 2010 Nov-Dec;16(6):745-60. doi: 10.1093/humupd/dmq011. Epub 2010 May 28. PMID 20511398
- [Background] Huser S, Guth S, Joost HG, Soukup ST, Kohrle J, Kreienbrock L, Diel P, Lachenmeier DW, Eisenbrand G, Vollmer G, Nothlings U, Marko D, Mally A, Grune T, Lehmann L, Steinberg P, Kulling SE. Effects of isoflavones on breast tissue and the thyroid hormone system in humans: a comprehensive safety evaluation. Arch Toxicol. 2018 Sep;92(9):2703-2748. doi: 10.1007/s00204-018-2279-8. Epub 2018 Aug 21. PMID 30132047
- [Background] Utian WH, Jones M, Setchell KD. S-equol: a potential nonhormonal agent for menopause-related symptom relief. J Womens Health (Larchmt). 2015 Mar;24(3):200-8. doi: 10.1089/jwh.2014.5006. Epub 2015 Feb 18. PMID 25692726
- [Background] Kim IS. Current Perspectives on the Beneficial Effects of Soybean Isoflavones and Their Metabolites for Humans. Antioxidants (Basel). 2021 Jun 30;10(7):1064. doi: 10.3390/antiox10071064. PMID 34209224
- [Background] Ishiwata N, Melby MK, Mizuno S, Watanabe S. New equol supplement for relieving menopausal symptoms: randomized, placebo-controlled trial of Japanese women. Menopause. 2009 Jan-Feb;16(1):141-8. doi: 10.1097/gme.0b013e31818379fa. PMID 19131846
- [Background] Aso T. Equol improves menopausal symptoms in Japanese women. J Nutr. 2010 Jul;140(7):1386S-9S. doi: 10.3945/jn.109.118307. Epub 2010 May 19. PMID 20484552
- [Background] Aso T, Uchiyama S, Matsumura Y, Taguchi M, Nozaki M, Takamatsu K, Ishizuka B, Kubota T, Mizunuma H, Ohta H. A natural S-equol supplement alleviates hot flushes and other menopausal symptoms in equol nonproducing postmenopausal Japanese women. J Womens Health (Larchmt). 2012 Jan;21(1):92-100. doi: 10.1089/jwh.2011.2753. Epub 2011 Oct 12. PMID 21992596
- [Background] Jenks BH, Iwashita S, Nakagawa Y, Ragland K, Lee J, Carson WH, Ueno T, Uchiyama S. A pilot study on the effects of S-equol compared to soy isoflavones on menopausal hot flash frequency. J Womens Health (Larchmt). 2012 Jun;21(6):674-82. doi: 10.1089/jwh.2011.3153. Epub 2012 Mar 12. PMID 22409590
- [Background] Setchell KD, Cole SJ. Method of defining equol-producer status and its frequency among vegetarians. J Nutr. 2006 Aug;136(8):2188-93. doi: 10.1093/jn/136.8.2188. PMID 16857839